CLINICAL TRIAL: NCT00850720
Title: Prevalence of Neuroendocrine Dysfunction in the Pediatric Cardiopulmonary Bypass Patient
Brief Title: Study of Possible Brain Hormone Problems After Open Heart Surgery in Infants
Status: Terminated | Type: Observational
Why Stopped: Inability to recruit / logistic problems.
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Kiran Hebbar, Assistant Professor - CT, Emory University
Other Study IDs: IRB00007443
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Results first posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Heart Disease
Keywords: Biological Response Modifiers; Bypass Surgery; Cardiology; Congenital Heart Disease; Endocrinology; Hormone Dysfunction; Hormones; Neuroendocrinology; Pediatric Surgery
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Blood Specimen Collection; Hydrocortisone; Arginine Vasopressin; Thyrotropin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Surgery: Infants with congenital defects.
  Interventions: Other: Blood draws

INTERVENTIONS:
Other: Blood draws — Samples of blood to be drawn before surgery, and nine hours after surgery.
  Other Names: Tests being analyzed:; • Cortisol; • Vasopressin (ADH); • Cortisol Free; • Thyroid Stimulating Hormone (TSH); • Free Thyroxine(FT4)

SUMMARY:
The goal of this study is to evaluate specific hormone levels in children undergoing heart surgery in order to identify patterns associated with any unstable vital signs. The data collected will provide preliminary answers to the question "Are hormone values a determining factor for drug administration and dosing levels?" and help establish the benefits of routine steroid and hormone administration. Sixty subjects will be enrolled. Blood samples will be drawn before the surgery,and again nine hours after surgery for analysis. Other patient data such as medications, vital signs, routine lab values and treatments will also be analyzed. As our current standard of care includes routine doses of steroids, we believe this study will increase our general knowledge and improve the care of these critically ill children. The study will also provide the foundation needed for grant support from the American Heart Association, allowing for future larger scale studies.

ELIGIBILITY:
Inclusion Criteria:

* Children with congenital heart disease requiring cardiopulmonary bypass(CPB) surgery less than 1 year of age admitted to the cardiac intensive care unit (CICU) preoperatively, who required blood sampling as part of their care.
* Subject must have arterial or central venous lines to be enrolled.
* Subject must have a documented weight of 2.5 Kilograms or greater.
* Subjects' legal guardian shall possess the ability to understand the purposes and risks of the study and provide an informed consent signature.

Exclusion Criteria:

* Medical urgency preventing timely administration of the consenting process.
* Any condition that, in the opinion of the attending physician, would place the patient at undue risk by participating. Specific conditions might include, but are not limited to, anemia or coagulopathy.
* Have given steroids intravenously (IV) or oral steroids within the last month.
* Have a preexisting neuroendocrine disorder.
* Have been treated with antipsychotic medication.
* Have human immunodeficiency virus (HIV).
* Have received etomidate for intubation.
* Other technical considerations that would prevent acquisition of sufficient samples OR inability / unwillingness of the legal guardian to provide consent.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients at Childrens Healthcare of Atlanta at Egleston
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2009-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Hebbar, MBBS, Principal Investigator — Emory University & Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiac Surgery
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Surgery
Number analyzed (Participants) | 0
Age, Categorical [Count of Participants; unit: Participants]
Age Continuous [Mean (Standard Deviation); unit: years]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: NO Outcomes - Study Terminated Without Data.
Time Frame: Study terminated - no data.
Arm/Group | Cardiac Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Cardiac Surgery
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Early termination of study; Technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes